CLINICAL TRIAL: NCT01700751
Title: A Pilot Study of Brentuximab Vedotin in the Prevention of Graft-Versus-Host Disease (GVHD) After Unrelated Allogeneic Stem Cell Transplantation
Brief Title: Brentuximab Vedotin Prevention of (GVHD) After Unrelated Allogeneic Stem Cell Transplantation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201211047
Record Dates: First submitted 2012-09-18; First posted 2012-10-04 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Leukemia, Acute Myeloid; Leukemia, Lymphoblastic,Acute; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose Level 0 (starting dose) (Experimental): brentuximab vedotin 0.3mg/kg, given IV on Days 7, 28, 49 & 70
  Interventions: Drug: brentuximab vedotin
- Dose Level 1 (Experimental): brentuximab vedotin 0.6mg/kg, given IV on Days 7, 28, 49 & 70
  Interventions: Drug: brentuximab vedotin
- Dose Level 2 (Experimental): brentuximab vedotin 1.2mg/kg, given IV on Days 7, 28, 49 & 70
  Interventions: Drug: brentuximab vedotin
- Dose Level 3 (Experimental): brentuximab vedotin 1.8mg/kg, given IV on Days 7, 28, 49 & 70
  Interventions: Drug: brentuximab vedotin
- Control Dose Level (No Intervention): The first 3 patients will not receive brentuximab vedotin.

INTERVENTIONS:
Drug: brentuximab vedotin
  Other Names: Adcetris
  Arms: Dose Level 0 (starting dose); Dose Level 1; Dose Level 2; Dose Level 3

SUMMARY:
This pilot clinical trial studies the safety and maximum tolerated dose of brentuximab vedotin when given with tacrolimus and methotrexate after unrelated allogeneic donor stem cell transplant in patients with acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndromes. The addition of brentuximab vedotin to tacrolimus and methotrexate may result in a significant reduction of graft versus host disease in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be scheduled to undergo stem cell transplantation for one of the following diagnoses:

  * acute myeloid leukemia (AML) in CR1 (first complete remission, CR or CRi) or CR2 (second complete remission, CR or CRi),
  * acute lymphoblastic leukemia (ALL) in CR1 or CR2 (CR or CRi)
  * myelodysplastic syndrome (MDS) without progression to AML.
  * Chronic myelogenous leukemia (CML)
  * Non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD)
  * Chronic lymphocytic leukemia (CLL)
  * Multiple myeloma (MM)
* Patients must be the recipient of unrelated donor peripheral blood stem cell products. Mismatches at both antigen and allele level will be eligible. Match must be 6 or 7 out of 8 loci (HLA A, B, C, and DRB1).
* Patient must receive any one of the following conditioning regimens: total body radiation (single or fractionated dose)/cyclophosphamide, busulfan/ cyclophosphamide, or fludarabine/busulfan/lymphocyte immune globulin (ATGAM/thymo).
* Patient must be ≥ 18 years and ≤ 70 years of age.
* Patient must have an ECOG performance status ≤ 2 or Karnofsky performance scale ≥ 60%
* Patient must have CD34+ stem cells ≥ 2x106/kg (actual body weight of the recipient) available for transplantation.
* Patient must have appropriate organ function as defined below (this criterion should be met on screening and on the day of the first dose of brentuximab vedotin (as assessed prior to dosing)):

  * Total bilirubin ≤ 2.0 x IULN
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x IULN
  * Serum creatinine ≤ 2.0 x IULN
  * Estimated Creatinine Clearance > 30 ml/min
  * Cardiac ejection fraction > 40%
  * DLCO/VA > 40%
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Patient must be able to understand and willing to sign an IRB approved written informed consent document.

Exclusion Criteria:

* Patient must not have had prior exposure to brentuximab vedotin.
* Patient must not have a history of other malignancy that has not been in remission for at least 3 years, with the exception of basal non-melanoma skin cancer which were treated with local resection only or intraepithelial lesions or carcinoma in situ of the cervix or prostate that has been curatively treated.
* Patient must not be receiving any other investigational agents.
* Patient must not have active CNS involvement.
* Patient must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to brentuximab vedotin or other agents used in the study.
* Patients must not have had previous radiation therapy to the mediastinum or lungs.
* Patient must not have an uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, active pulmonary diseases, or psychiatric illness/social situations that would limit compliance with study requirements (this criterion should be met on screening and on the day of but prior to first dose of brentuximab vedotin).
* Patient must not be pregnant and/or breastfeeding.
* Patient must not be known to be HIV-positive on combination antiretroviral therapies.
* Patient must not have had a previous allogeneic or syngeneic transplant. Prior autologous transplant is allowed.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-02-25 (Actual); Primary Completion 2015-11-11 (Actual); Study Completion 2016-11-21 (Actual)

PRIMARY OUTCOMES:
MTD of brentuximab vedotin when administered with a GVHD prophylaxis regimen | 37 days
  Defined as the dose level immediately below the dose level at which 2 patients of a cohort (of 2 to 6 patients) experience dose-limiting toxicity; Hematologic DLT is defined as ANC < 500/mm3 for three consecutive days beyond Day +21 that was determined by the investigator to be likely related to brentuximab vedotin.
  Non-hematologic DLT is defined as any grade 3 or higher non-hematologic toxicity that was determined by the investigator to be possibly, probably, or definitely related to brentuximab vedotin, with the following specific exceptions:
  * Grade 3 or 4 nausea, vomiting, diarrhea, mucositis, or fatigue thought to be associated with conditioning regimens
  * Grade 3 rash will only be considered a DLT for patients who have received two weeks of supportive care treatment with no improvement.

SECONDARY OUTCOMES:
Safety and tolerability of brentuximab vedotin when administered with a GVHD prophylaxis regimen | 100 days
  Toxicities described and graded using CTCAE version 4.0; described by patient, type, and grade for each dose level; summarized by counts and percentage of patients in the corresponding categories
Rate of acute GVHD | 100 days
  Proportion of all subjects who experience symptoms consistent with grade 2-4 acute GVHD; using the standard grading system adapted from the Glucksberg clinical stage and grade of acute GVHD
Rate of chronic GVHD | 2 years
  Proportion of all subjects who experience symptoms consistent with chronic GVHD; assessment will begin after Day 100 using the NIH consensus criteria for diagnosis and staging of chronic GVHD
Progression-free survival | 2 years
  Duration from the time of transplant to time of first progression, death, relapse after complete response, or the date the patient was last known to be in remission; estimated with Kaplan-Meier methods.
Overall survival. | 2 years
  Duration from the time of transplant to death or last follow-up; estimated with Kaplan-Meier methods.
1-year non-relapse mortality rate | 1 year
  Defined as the percentage of patients dying from etiologies other than disease relapse; estimated with Kaplan-Meier methods.
2-year non-relapse mortality rate | 2 years
  Defined as the percentage of patients dying from etiologies other than disease relapse; estimated with Kaplan-Meier methods.
1-year disease relapse rate | 1 year
  Defined as the percentage of patients who have disease relapse; estimated with Kaplan-Meier methods.
2-year disease relapse rate | 2 years
  Defined as the percentage of patients who have disease relapse; estimated with Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Schroeder, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu